CLINICAL TRIAL: NCT00180661
Title: Inflammation and Corticosteroid Responsiveness in Severe Asthma
Acronym: SARP
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Fan Chung, Professor, Imperial College London
Other Study IDs: HL-69155
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Results first posted 2019-10-04 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Asthma
Keywords: Severe asthma; corticosteroid responsiveness
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — endobronchial biopsies and blood specimens.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Severe Asthma: Patients under Steps 4/5 of Asthma Treatment - SIGN/BTS Guidelines
- Moderate Asthma: Asthma patients on steps 2/3 of Asthma treatment according to SIGN/BTS Guidelines
- Mild Asthma: Asthma patients on steps 1 of asthma treatment (steroid naive).

SUMMARY:
Some patients with mild asthma may develop severe asthma. It is not known what makes patients with mild asthma become severe, and we plan to find out why this happens. Patients with severe asthma may have a different type of inflammation in the airway tubes. Patients with severe asthma do not get as much benefit from taking steroid inhalers or tablets compared to asthma patients with mild disease. The study hypothesis is that the inflammation in severe asthma is such that it makes steroids less effective in treating asthma. We will find out what possible abnormalities there are in the blood cells and the bronchoalveolar macrophage cells in the lungs of patients with severe asthma compared to those with mild or moderate asthma.

DETAILED DESCRIPTION:
Study Design Patients referred to the Royal Brompton Hospital with severe asthma will be entered into a protocol that will determine whether they have asthma, and if so, the severity and clinical features of their asthma. Patients will also undergo investigations relating to asthma as detailed below. We will use an agreed Severe Asthma Research protocol (SARP) screening system to diagnose asthma (history, bronchodilator response and presence of bronchial hyperresponsiveness) (Screening questionnaire in SARP Handbook). Usually, the protocol will be carried out while the patient is admitted over 3-night admission.

Patients will undergo fiberoptic bronchoscopy. We will obtain cells by bronchoalveolar lavage and bronchial biopsies of the airway mucosa. These cells and biopsies will be studied in vitro as to the expression of corticosteroid receptor nuclear translocation, expression of cytokines, and the degree of histone acetylation/deacetylation status. These findings will be compared to those cells and biopsies obtained from mild and moderately severe asthma.

In a subgroup of patients with severe asthma, patients will be treated with oral prednisolone 40 mg/day or increase in maintenance dose of prednisolone by 40 mg/day. Fiberoptic bronchoscopy will then be repeated.

Details of the interventions proposed Some of the interventions listed below are in routine clinical use for investigation of severe asthma. For example, the computed tomogram is only ordered on clinical grounds. A fiberoptic bronchoscopy will be performed.

1. Demographic history and history of their symptoms of asthma and treatments using a comprehensive questionnaire
2. Quality of life questionnaire (AQLQ)
3. Skin prick tests to 16 common allergens
4. Measuring lung function tests
5. Bronchial responsiveness to methacholine
6. Bronchial reversibility test to inhaled salbutamol
7. Keeping a diary card of symptoms, treatments and peak flows for 2 weeks
8. Observance of compliance to treatments
9. Provision of sample of sputum, spontaneous or induced
10. Measuring exhaled nitric oxide; collecting of exhaled breath condensates
11. Fiberoptic bronchoscopy to obtain bronchoalveolar lavage cells, bronchial brushings and bronchial biopsies
12. Obtaining sample of blood for DNA extraction for genetic analysis
13. Obtaining blood for blood mononuclear cells for in vitro analysis of the effects of corticosteroids In patients with mild-to-moderate asthma, test 8 will not be performed. The details of these interventions are enclosed in the SARP Handbook.

Sources and Recruitment of Subjects:

Patients will be recruited from all patients referred to the Royal Brompton Hospital with a referral diagnosis of severe or difficult asthma for further management. The Royal Brompton Hospital is recognized nationally as a center for referral of such patients.

7Inclusion criteria The final diagnosis of severe asthma will be made according to the screening steps we have set up. The definition will require the presence of one or both major criteria (treatment with continuous or near continuous oral corticosteroids and/or requirement for treatment with high dose inhaled steroids) and two minor criteria.

Patients who do not fit the criteria of severe asthma will not be entered into the study.

Age 18-60; both sexes.

For the investigation of fiberoptic bronchoscopy, other additional inclusion criteria will be imposed:

1. Post-bronchodilator FEV1 greater than 40% on the day of the bronchoscopy
2. No evidence of an exacerbation of asthma within the past 4 weeks.
3. Ability to cooperate with procedures
4. Ability to give consent
5. The bronchoscopist has determined the subject is clinically appropriate for bronchoscopy

Patients will be excluded for fiberoptic bronchoscopy if:

1. FEV1 is less than 35% predicted before or less than 40% predicted after bronchodilator administration
2. Asthma is clinically unstable
3. Communication channels is not established for follow-up contacts
4. Clinically significant, unstable co-morbidities are present

Exclusion criteria Current smokers, and ex-smokers with greater than 10 pack years history of smoking.

Pregnancy or unreliable contraceptive measures in child-bearing woman.

Volunteer subjects We will need comparative asthmatic subjects with mild to moderately severe asthma. The groups will be defined as follows, according to their need for treatments (as established in the Asthma Management GINA or BTS guidelines): (i) Mild: intermittent symptoms and need for reliever bronchodilator less than once a day; (ii) moderate asthma: well-controlled asthma with minimal symptoms while on inhaled corticosteroid therapy not exceeding 2,000 microgram beclomethasone equivalent .

These patients will be recruited from the Asthma clinics attending the Royal Brompton Hospital, and also the milder patients will be recruited by advertisement within the Hospital, or from local general practices.

Current involvement in research The patients entered into this study will not be involved in any other research project, and must have Completed any other project within a month of entry into the current study. From previous experience, we aim to recruit 12 patients with severe asthma per year; in total, 50 patients with severe asthma over a 4 year period. Concomitantly, we will recruit 40 mild-to-moderately severe asthma patients. Pharmacology and Dispensing (i) substance: Prednisolone tablets (ii) route of administration: Oral (iii) frequency : once a day (iv) dosage: 30 mg/day (or addition of 30 mg on top of maintainence dose) (v) stage of CSM evaluation: n/a.

ELIGIBILITY:
Inclusion Criteria:

The final diagnosis of severe asthma will be made according to the screening steps we have set up. The definition will require the presence of one or both major criteria (treatment with continuous or near continuous oral corticosteroids and/or requirement for treatment with high dose inhaled steroids) and two minor criteria.

Patients who do not fit the criteria of severe asthma will not be entered into the study.

Age 18-60; both sexes.

For the investigation of fiberoptic bronchoscopy, other additional inclusion criteria will be imposed:

1. Post-bronchodilator FEV1 greater than 40% on the day of the bronchoscopy
2. No evidence of an exacerbation of asthma within the past 4 weeks.
3. Ability to cooperate with procedures
4. Ability to give consent
5. Current smokers, and ex-smokers with greater than 10 pack years history of smoking.

Exclusion criteria

Pregnancy or unreliable contraceptive measures in child-bearing woman. he bronchoscopist has determined the subject is clinically appropriate for bronchoscopy

-

Exclusion Criteria:

-

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Asthma population living in the UK - ranging in severity (from mild, to severe).
Sampling Method: Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2003-08 (Actual); Primary Completion 2008-02 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kian Fan Chung, MD, Principal Investigator — Imperial College London
Locations (1):
- Royal Brompton Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chung KF, Godard P, Adelroth E, Ayres J, Barnes N, Barnes P, Bel E, Burney P, Chanez P, Connett G, Corrigan C, de Blic J, Fabbri L, Holgate ST, Ind P, Joos G, Kerstjens H, Leuenberger P, Lofdahl CG, McKenzie S, Magnussen H, Postma D, Saetta M, Salmeron S, Sterk P. Difficult/therapy-resistant asthma: the need for an integrated approach to define clinical phenotypes, evaluate risk factors, understand pathophysiology and find novel therapies. ERS Task Force on Difficult/Therapy-Resistant Asthma. European Respiratory Society. Eur Respir J. 1999 May;13(5):1198-208. doi: 10.1034/j.1399-3003.1999.13e43.x. No abstract available. PMID 10414427
- [Result] Bhavsar P, Hew M, Khorasani N, Torrego A, Barnes PJ, Adcock I, Chung KF. Relative corticosteroid insensitivity of alveolar macrophages in severe asthma compared with non-severe asthma. Thorax. 2008 Sep;63(9):784-90. doi: 10.1136/thx.2007.090027. Epub 2008 May 20. PMID 18492738

RESULTS

PARTICIPANT FLOW:
Groups:
- Non-severe Asthma: Patients with Non-severe asthma
- Severe Asthma: Patients with severe asthma
Period: Overall Study
Arm/Group | Non-severe Asthma | Severe Asthma
Started | 19 | 20
Completed | 19 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Non-severe Asthma | Severe Asthma | Total
Number analyzed (Participants) | 19 | 20 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (2.4) | 41.4 (2.6) | 40.7 (2.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 14 | 21
  Male | 12 | 6 | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 19 | 20 | 39

OUTCOME MEASURES:

1. Primary Outcome: Lung Function FEV1
Description: FEV1, or forced expiratory volume, is a measurement taken from a pulmonary function test. It calculates the amount of air that a person can force out of their lungs in 1 second.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: % of predicted
Arm/Group | Non-severe Asthma | Severe Asthma
Number analyzed (Participants) | 19 | 20
% of predicted | 84.9 (3) | 59.9 (4.4)
Statistical Analysis 1: Comparison: Non-severe Asthma vs Severe Asthma; Test type: Superiority; p = 0.001, t-test, 2 sided

2. Primary Outcome: Suppression of Monocyte Activation and Alveolar Macrophage Activation by Dexamethasone Ex-vivo
Description: IL8 - Interleukin-8 (IL-8) is a cytokine produced by many normal cells including monocytes, neutrophils, fibroblasts, and endothelial cells
Time Frame: 1 day
Measure: Mean (Full Range); unit: % of supression
Arm/Group | Non-severe Asthma | Severe Asthma
Number analyzed (Participants) | 19 | 20
% of supression | 30 [25 to 75] | 10 [5 to 10]
Statistical Analysis 1: Comparison: Non-severe Asthma vs Severe Asthma; Test type: Superiority; p = 0.005, t-test, 2 sided

3. Primary Outcome: Effect of Corticosteroids on Release of Cytokines From Macrophages
Time Frame: Once
Population: No data collected
Arm/Group | Non-severe Asthma | Severe Asthma
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Exhaled NO
Time Frame: 1 day
Population: No data collected
Arm/Group | Non-severe Asthma | Severe Asthma
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Biopsy Eosinophils
Time Frame: Once
Population: No data collected
Arm/Group | Non-severe Asthma | Severe Asthma
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Sputum Eosinophils
Time Frame: Once
Population: No data collected
Arm/Group | Non-severe Asthma | Severe Asthma
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Non-severe Asthma | Severe Asthma
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/20
Other Adverse Events (participants affected / at risk) | 0/19 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes